CLINICAL TRIAL: NCT01773187
Title: A Randomized Controlled Phase 3 Study of Oral Pacritinib Versus Best Available Therapy in Patients With Primary Myelofibrosis, Post-Polycythemia Vera Myelofibrosis, or Post-Essential Thrombocythemia Myelofibrosis
Brief Title: Pacritinib Versus Best Available Therapy to Treat Myelofibrosis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PERSIST-1 (PAC325)
Record Dates: First submitted 2013-01-18; First posted 2013-01-23 (Estimated); Results first posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Primary Myelofibrosis; Post-polycythemia Vera Myelofibrosis; Post-essential Thrombocythemia Myelofibrosis
Keywords: Myelofibrosis; Post-Polycythemia Vera Myelofibrosis; Post-Essential Thrombocythemia Myelofibrosis; Primary Myelofibrosis; Polycythemia Vera; Essential Thrombocythemia; Bone Marrow Disease; Hematologic Disease; Splenomegaly; Pacritinib; MPN-SAF; MPN-SAF TSS; Anemia; Myeloproliferative Neoplasm; Spleen volume; Thrombocytopenia; SB1518
MeSH Terms: conditions — Primary Myelofibrosis; Polycythemia Vera; Thrombocythemia, Essential; Bone Marrow Diseases; Hematologic Diseases; Splenomegaly; Anemia; Myeloproliferative Disorders; Thrombocytopenia | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pacritinib (Experimental): Pacritinib 400 mg QD
  Interventions: Drug: Pacritinib
- Best Available Therapy (Active Comparator): BAT includes any physician-selected treatment for primary or secondary myelofibrosis with the exclusion of JAK inhibitors (inhibitors of Janus kinases)
  Interventions: Drug: Best Available Therapy

INTERVENTIONS:
Drug: Pacritinib
  Arms: Pacritinib
Drug: Best Available Therapy
  Arms: Best Available Therapy

SUMMARY:
Phase 3, randomized, controlled study to evaluate the safety and efficacy of oral pacritinib compared to Best Available Therapy (BAT) in patients with primary or secondary myelofibrosis.

DETAILED DESCRIPTION:
Multicenter, randomized, controlled, phase 3 trial comparing the safety and efficacy of pacritinib with that of BAT in patients with primary or secondary myelofibrosis. Approximately 322 eligible patients will be randomized in a 2:1 allocation to pacritinib (400mg QD) or BAT (includes any physician-selected treatment for myelofibrosis with the exclusion of JAK inhibitors (inhibitors of Janus kinases)). Spleen volume will be measured by MRI or CT at baseline and every 12 weeks thereafter. An independent radiology facility (IRF), blind to treatment assignments, will measure spleen volumes. Patients will also be followed for safety, Leukemia Free Survival (LFS), Overall Survival (OS), frequency of red blood cell (RBC) and platelet transfusions, and other exploratory endpoints. An Independent Data Monitoring Committee (IDMC) will evaluate the safety of pacritinib.

ELIGIBILITY:
Inclusion Criteria:

* Intermediate -1 or -2 or high-risk Myelofibrosis (per Passamonti et al 2010)
* Palpable splenomegaly ≥ 5 cm on physical examination
* Total Symptom Score >13 on the MPN-SAF TSS 2.0, not including the inactivity question
* Patients who are platelet or red blood cell transfusion-dependent are eligible
* Adequate white blood cell counts (with low blast counts), liver function, and renal function
* No spleen radiation therapy for 6-12 months
* Last therapy for myelofibrosis was 2-4 weeks ago, including any erythropoietic or thrombopoietic agent
* Not pregnant, not lactating, and agree to use effective birth control

Exclusion Criteria:

* Prior treatment with a JAK2 inhibitor
* History of (or plans to undergo) spleen removal surgery or allogeneic stem cell transplant
* Ongoing gastrointestinal medical condition such as Crohn's disease, Inflammatory bowel disease, chronic diarrhea, or constipation
* Cardiovascular disease, including recent history or currently clinically symptomatic and uncontrolled: congestive heart failure, arrhythmia, angina, QTc prolongation or other QTc risk factors, myocardial infarction
* Other malignancy within last 3 years other than certain limited skin, cervical, prostate, breast, or bladder cancers
* Other ongoing, uncontrolled illnesses (including HIV infection and active hepatitis A, B, or C), psychiatric disorder, or social situation that would prevent good care on this study
* Life expectancy < 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth Ziemba, Study Director — VP, Pharmacovigilance, Clinical Operations, QA
Locations (81):
- United States (4):
  - CTI Investigational Site 10002, Scottsdale, Arizona
  - CTI Investigational Site 10004, Omaha, Nebraska
  - CTI Investigational Site 10001, Morristown, New Jersey
  - CTI Investigational Site 10003, Greenville, South Carolina
- Australia (6):
  - CTI Investigational Site 61006, Box Hill
  - CTI Investigational Site 61001, Coffs Harbour
  - CTI Investigational Site 61005, Geelong
  - CTI Investigational Site 61003, Gosford
  - CTI Investigational Site 61004, Hobart
  - CTI Investigational Site 61002, Milton
- Belgium (5):
  - CTI Investigational Site 32002, Antwerp
  - CTI Investigational Site 32003, Antwerp
  - CTI Investigational Site 32001, Bruges
  - CTI Investigational Site 32005, Brussels
  - CTI Investigational Site 32004, La Louvière
- Czechia (4):
  - CTI Investigational Site 42003, Brno
  - CTI Investigational Site 42001, Olomouc
  - CTI Investigational Site 42002, Pilsen
  - CTI Investigational Site 42004, Prague
- France (12):
  - CTI Investigational Site 33005, Amiens
  - CTI Investigational Site 33006, Caen
  - CTI Investigational Site 33011, Grenoble
  - CTI Investigational Site 33012, Lens
  - CTI Investigational Site 33007, Lille
  - CTI Investigational Site 33001, Nîmes
  - CTI Investigational Site 33004, Paris
  - CTI Investigational Site 33008, Paris
  - CTI Investigational Site 33009, Pessac
  - CTI Investigational Site 33010, Pierre-Bénite
  - CTI Investigational Site 33003, Strasbourg
  - CTI Investigational Site 33002, Toulouse
- Germany (9):
  - CTI Investigational Site 49006, Berlin
  - CTI Investigational Site 49007, Berlin
  - CTI Investigational Site 49001, Cologne
  - CTI Investigational Site 49003, Dresden
  - CTI Investigational Site 49008, Essen
  - CTI Investigational Site 49002, Freiburg im Breisgau
  - CTI Investigational Site 49005, Mainz
  - CTI Investigational Site 49004, München
  - CTI Investigational Site 49009, Münster
- Hungary (8):
  - CTI Investigational Site 36002, Budapest
  - CTI Investigational Site 36005, Debrecen
  - CTI Investigational Site 36006, Gyula
  - CTI Investigational Site 36003, Kaposvár
  - CTI Investigational Site 36004, Kecskemét
  - CTI Investigational Site 36001, Szeged
  - CTI Investigational Site 36008, Szolnok
  - CTI Investigational Site 36007, Szombathely
- Italy (7):
  - CTI Investigational Site 39003, Bologna
  - CTI Investigational Site 39001, Florence
  - CTI Investigational Site 39005, Milan
  - CTI Investigational Site 39004, Monza
  - CTI Investigational Site 39002, Padua
  - CTI Investigational Site 39008, Reggio Emilia
  - CTI Investigational Site 39006, Rimini
- Netherlands (4):
  - CTI Investigational Site 31001, Amsterdam
  - CTI Investigational Site 31002, Maastricht
  - CTI Investigational Site 31003, Rotterdam
  - CTI Investigational Site 31004, Utrecht
- New Zealand (4):
  - CTI Investigational Site 64001, Christchurch
  - CTI Investigational Site 64004, Dunedin
  - CTI Investigational Site 64002, Hamilton
  - CTI Investigational Site 64003, Takapuna
- Russia (10):
  - CTI Investigational Site 70011, Izhevsk
  - CTI Investigational Site 70008, Moscow
  - CTI Investigational Site 70009, Moscow
  - CTI Investigational Site 70002, Petrozavodsk
  - CTI Investigational Site 70001, Saint Petersburg
  - CTI Investigational Site 70004, Saint Petersburg
  - CTI Investigational Site 70010, Saint Petersburg
  - CTI Investigational Site 70005, Samara
  - CTI Investigational Site 70006, Sochi
  - CTI Investigational Site 70007, Volgograd
- United Kingdom (8):
  - CTI Investigational Site 44004, Birmingham
  - CTI Investigational Site 44008, Bournemouth
  - CTI Investigational Site 44002, Cambridge
  - CTI Investigational Site 44003, Cardiff
  - CTI Investigational Site 44001, London
  - CTI Investigational Site 44007, London
  - CTI Investigational Site 44006, Manchester
  - CTI Investigational Site 44005, Oxford

REFERENCES:
- [Background] Mesa RA, Vannucchi AM, Mead A, Egyed M, Szoke A, Suvorov A, Jakucs J, Perkins A, Prasad R, Mayer J, Demeter J, Ganly P, Singer JW, Zhou H, Dean JP, Te Boekhorst PA, Nangalia J, Kiladjian JJ, Harrison CN. Pacritinib versus best available therapy for the treatment of myelofibrosis irrespective of baseline cytopenias (PERSIST-1): an international, randomised, phase 3 trial. Lancet Haematol. 2017 May;4(5):e225-e236. doi: 10.1016/S2352-3026(17)30027-3. Epub 2017 Mar 20. PMID 28336242
- [Derived] Tremblay D, Mesa R, Scott B, Buckley S, Roman-Torres K, Verstovsek S, Mascarenhas J. Pacritinib demonstrates spleen volume reduction in patients with myelofibrosis independent of JAK2V617F allele burden. Blood Adv. 2020 Dec 8;4(23):5929-5935. doi: 10.1182/bloodadvances.2020002970. PMID 33275766

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pacritinib | Best Available Therapy
Started | 220 | 107
Completed | 167 | 75
Not Completed | 53 | 32

BASELINE CHARACTERISTICS:
Population: Represents Intent To Treat population (number of randomized patients)
Groups:
- Total: Total of all reporting groups
Arm/Group | Pacritinib | Best Available Therapy | Total
Number analyzed (Participants) | 220 | 107 | 327
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 85 | 52 | 137
  >=65 years | 135 | 55 | 190
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (10.85) | 64.8 (9.12) | 65.3 (10.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 47 | 142
  Male | 125 | 60 | 185
Region of Enrollment [Number; unit: participants]
  New Zealand | 16 | 4 | 20
  Netherlands | 13 | 8 | 21
  Belgium | 8 | 1 | 9
  Hungary | 49 | 21 | 70
  Czechia | 9 | 9 | 18
  United States | 3 | 2 | 5
  Italy | 11 | 10 | 21
  United Kingdom | 19 | 6 | 25
  Australia | 29 | 17 | 46
  France | 26 | 9 | 35
  Germany | 2 | 2 | 4
  Russia | 35 | 18 | 53

OUTCOME MEASURES:

1. Primary Outcome: Spleen Volume Reduction
Description: Number of patients achieving a ≥ 35% reduction in spleen volume from baseline to week 24 as measured by magnetic resonance imaging (MRI) or computed tomography (CT)
Time Frame: Baseline to Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Pacritinib | Best Available Therapy
Number analyzed (Participants) | 220 | 107
Participants | 42 | 5
Statistical Analysis 1: Comparison: Pacritinib vs Best Available Therapy; Pre-specified; Test type: Superiority; p = 0.0003, Fisher Exact

2. Secondary Outcome: Total Symptom Score (TSS) Reduction
Description: Number of patients with >= 50% reduction in total score from baseline to week 24 on the Myeloproliferative Neoplasm Symptom Assessment Form 2.0 (MPN-SAF TSS 2.0). Responses (on a scale from 0 [absent] to 10 [worst imaginable]) to questions about symptoms (tiredness, early satiety, abdominal discomfort, night sweats, pruritus, bone pain, and pain under the ribs on the left side) were used to calculate the TSS.
Time Frame: Baseline to Week 24
Population: The original version (MPN-SAF TSS) was administered to the first 179 subjects enrolled in the study. The subsequent 148 enrolled subjects were administered the MPN-SAF TSS 2.0 and comprise the ITT population for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Pacritinib | Best Available Therapy
Number analyzed (Participants) | 100 | 48
Participants | 19 | 5
Statistical Analysis 1: Comparison: Pacritinib vs Best Available Therapy; Pre-specified; Test type: Superiority; p = 0.2368, Fisher Exact

ADVERSE EVENTS:
Time Frame: Time of signing informed consent through 30 days after the last study treatment.
Description: The data display threshold for SAEs is set to 1% or more, that of AEs is set to 5% or more.
Arm/Group | Pacritinib | Best Available Therapy
All-Cause Mortality (participants affected / at risk) | 27/220 | 3/106
Serious Adverse Events (participants affected / at risk) | 117/220 | 33/106
Other Adverse Events (participants affected / at risk) | 207/220 | 81/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pacritinib (N=220) | Best Available Therapy (N=106)
Basal cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 2 (2)
Squarmous cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (10) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (7) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 4 (6) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
Anemia (Blood and lymphatic system disorders) | 16 (20) | 5 (106)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 (4) | 0 (0)
Disease Progression (General disorders) | 6 (6) | 3 (3)
Pyrexia (General disorders) | 6 (6) | 3 (4)
Multi-organ failure (General disorders) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 4 (4) | 0 (0)
Pneumonia (Infections and infestations) | 16 (21) | 4 (4)
Lobar pneumonia (Infections and infestations) | 4 (4) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 3 (3) | 1 (1)
Sepis (Infections and infestations) | 2 (3) | 2 (2)
Cardiac Failure (Cardiac disorders) | 7 (7) | 3 (3)
Clonal evolution (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Epstein-Barr virus associated lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pacritinib (N=220) | Best Available Therapy (N=106)
Hypertension (Vascular disorders) | 11 (11) | 0 (0)
Fatigue (General disorders) | 33 (33) | 9 (9)
Oedema peripheral (General disorders) | 24 (24) | 16 (16)
Pyrexia (General disorders) | 17 (17) | 11 (11)
Asthernia (General disorders) | 16 (16) | 7 (7)
Insomnia (Psychiatric disorders) | 13 (13) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 11 (11) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 12 (12) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 58 (58) | 18 (18)
Thrombocytopenia (Blood and lymphatic system disorders) | 48 (48) | 15 (15)
Neutropenia (Blood and lymphatic system disorders) | 12 (12) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 (20) | 9 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 10 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 8 (8)
Oropharyngeal (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 0 (0)
Headache (Nervous system disorders) | 12 (12) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 142 (142) | 14 (14)
Nausea (Gastrointestinal disorders) | 70 (70) | 7 (7)
Vomiting (Gastrointestinal disorders) | 46 (46) | 7 (7)
Abdominal pain (Gastrointestinal disorders) | 29 (29) | 11 (11)
Constipation (Gastrointestinal disorders) | 22 (22) | 8 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 14 (14) | 0 (0)
Rush (Skin and subcutaneous tissue disorders) | 12 (12) | 0 (0)
Arthralgia (Skin and subcutaneous tissue disorders) | 13 (13) | 0 (0)
Pain in extremity (Skin and subcutaneous tissue disorders) | 11 (11) | 9 (9)
Decreased appetite (Metabolism and nutrition disorders) | 21 (21) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 16 (16) | 6 (6)
Urinary tract infection (Infections and infestations) | 12 (12) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other